CLINICAL TRIAL: NCT02495623
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multi-Dose Study of the Effect of Two Dosage Strengths of SYN-010 Compared With Placebo on Breath Methane Production in Breath Methane-Positive Subjects With IBS-C
Brief Title: A Study of the Effect of SYN-010 on Subjects With IBS-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theriva Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB-2-010-001
Record Dates: First submitted 2015-06-29; First posted 2015-07-13 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Active Comparator): 21 mg SYN-010
  Interventions: Drug: SYN-010 21 mg
- High Dose (Active Comparator): 42 mg SYN-010
  Interventions: Drug: SYN-010 42 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYN-010 21 mg
  Arms: Low Dose
Drug: SYN-010 42 mg
  Arms: High Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multi-Dose Study of the Effect of Two Dosage Strengths of SYN-010 Compared with Placebo on Breath Methane Production in Breath Methane-Positive Subjects with Irritable Bowel Syndrome with Constipation (IBS-C)

DETAILED DESCRIPTION:
This is a Phase 2, randomized, multi-center, multi-dose study. Sixty subjects with irritable bowel syndrome with constipation who are between the ages of 18 and 65, inclusive, will be enrolled. The entire duration of the study may be up to 43 days (from Screening to the post end-of-study [EOS] visit telephone call).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have IBS-C and have a positive breath CH4 test result (> 10 ppm) at Screening.
* Subject must meet the modified Rome III criteria for IBS-C.
* Subject must have an average abdominal pain intensity score of ≥ 3 (scale 0-10) reported at Screening and Baseline.
* Subject must have an average of fewer than 3 complete spontaneous bowel movement (CSBMs) per week.
* Subject must agree to refrain from making any lifestyle changes that may affect IBS-C symptoms from the time of Screening to the end of the study.

Exclusion Criteria:

* Subject has taken IBS treatments (prescription or over-the-counter), proton pump inhibitors, laxatives, antibiotics.
* Subject currently has any structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility, or any unexplained and clinically significant symptoms such as lower GI bleeding, rectal bleeding, heme-positive stool, iron-deficiency anemia, weight loss, or systemic signs of infection.
* Subject has been diagnosed with or has a family history of familial adenomatous polyposis, hereditary nonpolyposis colorectal cancer, or any other form of familial colorectal cancer.
* Subject reports loose (mushy) or watery stools (Bristol Stool Form Scale [BSFS] score of 6 or 7).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kaleko, M.D., Study Director — Synthetic Biologics
Locations (1):
- Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 79 subjects were randomized into the study per IVRS. 63 subjects received at least one dose of SYN-010. 16/79 subjects were not administered a single dose of study drug or placebo. We considered the subject truly randomized once the subject had completed the breath methane test, completed the daily diary entries, and were assigned study drug.
Period: Overall Study
Arm/Group | Low Dose | High Dose | Placebo
Started | 25 | 26 | 28
Dosed | 22 | 19 | 22
Completed | 20 | 17 | 20
Not Completed | 5 | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 22 | 19 | 22 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (6.01) | 44.7 (9.54) | 46.4 (10.29) | 44.6 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 17 | 50
  Male | 3 | 5 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Area Under the Curve (AUC) of Breath CH4 Production at Day 7
Time Frame: 7 days
Population: 79 subjects consented/randomized to treatment. 63 dosed subjects. 59 subjects (21, 20 & 18 for the placebo, 21mg and 42mg, respectively) were included for the analysis of AUC on Day 7, and the subjects with missing CH4 values at either baseline or Day 7 were excluded from the analysis since the area under the curve could not be calculated.
Measure: Mean (Standard Deviation); unit: hours*ppm
Groups:
- Low Dose: 21 mg SYN-010
  SYN-010 21 mg
- High Dose: 42 mg SYN-010
  SYN-010 42 mg
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 20 | 18 | 21
hours*ppm | 99.2 (79.4) | 57.3 (43.1) | 72.7 (53.5)

ADVERSE EVENTS:
Arm/Group | Low Dose | High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 2/22 | 2/19 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=22) | High Dose (N=19) | Placebo (N=22)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
AST increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood CPK increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators do not see trial results ahead of public disclosure unless it is under CDA. Investigators will not be allowed to publish or disclose any study results prior to sponsor communicating it to the public.